CLINICAL TRIAL: NCT04983732
Title: A Randomized, Open-Label, Parallel Study to Evaluate the Absolute Bioavailability of FL-101 in Healthy Male and Female Subjects
Brief Title: A Bioavailability Study of FL-101 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flame Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL-101-1001
Record Dates: First submitted 2021-07-22; First posted 2021-07-30 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Healthy Subjects
Keywords: Absolute Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FL-101-IV (Experimental): FL-101 single IV infusion over 60-minutes
  Interventions: Drug: FL-101-Intravenous
- FL-101-SC (Experimental): FL-101 single SC injection
  Interventions: Drug: FL-101-Subcutaneous

INTERVENTIONS:
Drug: FL-101-Intravenous — 150 mg administered via the IV route
  Arms: FL-101-IV
Drug: FL-101-Subcutaneous — 150 mg administered via the SC route
  Arms: FL-101-SC

SUMMARY:
This will be a single-center, randomized, open-label, single dose, parallel study to assess the absolute bioavailability of FL-101 when administered via the subcutaneous (SC) and intravenous (IV) routes.

DETAILED DESCRIPTION:
This single-center, randomized, open-label, single dose, parallel study will assess the absolute bioavailability of 150 mg FL-101 when administered via the SC and IV routes. The study will consist of a Screening Period (up to 28 days), followed by Baseline assessments and an inpatient Study Treatment Period of 24 hours (Day 1 and Day 2). Subjects will return to the clinic as outpatients for study procedures including, but not limited to, blood samples to be obtained for both PK and antibody assessments at pre-specified time points.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between the ages of 18 and 55 years, inclusive, at Screening.
2. Willing and able to provide written informed consent prior to participating in the study.
3. Able to communicate clearly with the Investigator and staff; able to read, and understand study procedures.
4. Able to complete all Screening period evaluations, stay in the clinical research facility for the duration of the inpatient portion of the study, and attend scheduled follow-up visits by videoconference or teleconference, and/or in-person as needed. In the case of neutropenia, subject must be willing and able to return for follow-up blood counts, including after EOS (Day 85) visit.
5. BMI between 18 and 32.49 kg/m2, inclusive, and body weight not less than 50 kg.
6. In good general health, free from clinically significant medical or psychiatric illness or disease (as determined by medical/surgical history, physical examination, weight, 12-lead ECG, and clinical laboratory tests).
7. Vital signs at Screening must be within the following ranges and stable (measured in semi-reclined position after at least 5 minutes of rest):

   * SBP ≥90 and ≤150 mmHg
   * DBP ≥50 and ≤95 mmHg
   * HR ≥45 and ≤100 beats per minute (bpm)
   * Note: If vital signs are out of range, the Investigator may obtain one additional reading, so that up to two consecutive assessments are made within 1 hour, and with the volunteer semi-reclined quietly during the 5 minutes preceding the assessment.
8. A 12-lead ECG consistent with normal cardiac conduction and function at Screening, including: HR between 45 and 100 bpm; QTcF interval ≤460 ms; QRS interval <120 ms; PR interval <220 ms; and morphology consistent with healthy cardiac conduction and function.
9. Nonsmoker within the previous 6 months (before Screening), and does not use tobacco containing, or nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, e-cigarettes, nicotine patch, or nicotine gum).
10. Has clinical chemistry, hematology, coagulation, and complete urinalysis (fasted for at least 6 hours) results at Screening and at admission within the reference range for the testing laboratory unless the out-of-range results are deemed not clinically significant by the Investigator and the Sponsor.
11. Has adequate renal function at Screening and at admission as evidenced by creatinine clearance ≥ 90 mL/min by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) estimation.
12. Has adequate hepatic function at Screening and at admission as evidenced by the following: total bilirubin ≤ upper limit of normal (ULN); aspartate aminotransferase (AST) ≤ ULN and alanine aminotransferase (ALT) ≤ ULN.
13. Has a negative urine drug screen result at Screening and at admission.
14. Male subjects who are non-sterilized must agree to be sexually abstinent or use double barrier contraception (e.g., condom and spermicide) for 3 months (90 days) after receiving the study drug.
15. Male subjects must agree to not donate sperm from Screening and at least 3 months (90 days) after receiving the study drug.
16. Female subjects must be surgically sterilized, post-menopausal as defined by 1 year with no menses or using an adequate means of birth control if pre-menopausal.

Exclusion Criteria:

1. Has a history of or current clinically significant medical illness including (but not limited to) pulmonary, cardiovascular, renal, coagulation disorders, lipid abnormalities, gastrointestinal, immunologic, endocrine, neurologic, psychiatric, or thromboembolic disease, metabolic disturbances, or any other current physical condition that the Investigator (or designee) considers should exclude the participant, or that could interfere with the interpretation of the study results.
2. Has any clinically significant medical condition, physical examination finding, ECG abnormality, or clinically significant abnormal value for clinical chemistry, hematology, coagulation, or urinalysis at Screening or at admission to the study center, as deemed appropriate by the Investigator (or designee).
3. History or presence of malignancy within the past 5 years, with the exception of adequately treated localized skin cancer (basal cell or squamous cell carcinoma), which is allowed.
4. Currently suffers from clinically significant systemic allergic disease, or has a history of significant drug allergies, including but not limited to:

   * A history of anaphylactic reaction
   * Allergic reaction due to any drug that led to significant morbidity
   * Known hypersensitivity to any component of the formulation of test article (FL-101).
5. Has donated or intends to donate blood or blood products or has had an acute loss of blood (>500 mL) during the 60 days before study drug administration (10 days for plasma donation) or intends to donate blood or blood products within 2 months after the completion of the study.
6. Has had an acute, clinically significant illness within 30 days prior to Day 1, or has had a recent febrile illness with an abnormal body temperature within 72 hours prior to admission.
7. Has a history within the past 24 months before Screening of drug abuse (defined as any illicit drug use), or a history of alcohol abuse (defined as alcohol consumption exceeding 14 units per week). One unit of alcohol equals 360 mL (12 oz.) of beer, 45 mL (1.5 oz.) of liquor, or 150 mL (5 oz.) of wine.
8. Has a positive test for drugs of abuse at Screening or alcohol 3 days prior to dosing or is unwilling to abstain from alcohol and drugs of abuse throughout the study.
9. Has a smoking history during the past 6 months before Screening. This includes the use of any nicotine-containing substances (e.g., nicotine patch or gum, chewing tobacco, e-cigarettes), or has a positive cotinine test at Screening, or is unwilling to abstain from these products for the duration of the study.
10. Has used any investigational compound or an experimental medical device, within 30 days prior to receiving the study drug.
11. If male, the subject intends to impregnate others, or donate sperm within 90 days (3 months) after receiving the study drug.
12. Has inadequate venous access for the required blood draws for the study.
13. Is unable to meet or perform study requirements, or has a known or suspected inability to comply with the study protocol.
14. Is unable or unwilling to eat provided food (e.g., vegetarian, kosher, lactose intolerant dietary requirements).
15. Is an immediate family member of the Investigator, or is an employee of the study center, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
16. Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study drug based on Principal Investigator judgment.
17. Use of any OTC medication (including nutritional or dietary supplements, herbal preparations, or vitamins) within 7 days prior to receiving the study drug until the end of study visit.
18. Use of any prescription medication (except hormonal contraception) from 14 days prior to receiving the study drug until the end-of-study visit.
19. Use of TNF-blocker within 30 days prior to receiving the study drug until 3 months (90 days) after receiving the study drug.
20. Receipt of live or attenuated vaccine within 30 days prior to receiving the study drug until 3 months (90 days) after receiving the study drug. Subjects may receive the COVID-19 vaccine but must wait 2 weeks after receiving the 2nd dose of the vaccine to be enrolled into the study.
21. Engagement in non-routine strenuous exercise from 48 hours prior to receiving the study drug until the end-of-study visit.
22. Consumption of xanthines from 48 hours prior to admission until the end of study visit. Subjects will be instructed not to consume any of the above products; however, allowance for an isolated single incidental consumption may be evaluated and approved by the study Investigator based on the potential for interaction with the study drug.
23. Has a positive test for HBsAg, HCV antibody, or HIV at Screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.
24. Female subjects who are pregnant or lactating.
25. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
FL-101 Absolute Bioavailability | Day 1 to Day 85
  To determine the absolute bioavailability of FL-101 administered as a single dose via subcutaneous (SC) administration relative to a single intravenous (IV) dose in healthy male and female subjects.

SECONDARY OUTCOMES:
Serum concentration of FL-101 | Day 1 to Day 85
  To characterize the PK of FL-101 administered via the SC and IV routes in healthy male and female subjects.
Incidence of adverse events | Day 1 to Day 85
  To evaluate the safety and tolerability of FL-101 administered SC and IV in healthy male and female subjects.

OTHER OUTCOMES:
FL-101 Antibodies | Day 1 (predose) and Days 8, 15, 22, 29, 43, 57, 71, and 85
  To determine the presence of antibodies to FL-101 following SC and IV administration.

CONTACTS AND LOCATIONS:
Overall Officials: Swarna Yadlapalli, MD, Principal Investigator — Axis Clinicals
Locations (1):
- Axis Clinicals, Dilworth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No